CLINICAL TRIAL: NCT03434041
Title: A Randomized, Double-blind, Multicenter Active-controlled Study to Evaluate the Efficacy, Pharmacokinetics, Safety and Tolerability of Flexible Doses of Intranasal Esketamine Plus an Oral Antidepressant in Adult Subjects With Treatment-resistant Depression
Brief Title: A Study to Evaluate the Efficacy, Pharmacokinetics, Safety and Tolerability of Flexible Doses of Intranasal Esketamine Plus an Oral Antidepressant in Adult Participants With Treatment-resistant Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108418; ESKETINTRD3006 (Other: Janssen Research & Development, LLC)
Expanded Access: NCT03829579 (Approved for marketing)
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Results first posted 2022-05-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Esketamine; Duloxetine Hydrochloride; Antidepressive Agents; Escitalopram; Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal Esketamine plus Oral Antidepressant (Experimental): Eligible participants will self-administer esketamine (56 mg or 84 mg) intranasally twice per week for 4 weeks as a flexible dose regimen in the Double-Blind Treatment Phase. All participants will start at a dose of 56 milligram (mg) on Day 1. The dose may be increased to 84 mg or maintained at 56 mg per investigator's discretion. In addition, participants will simultaneously initiate a new, open-label 1 of 4 oral antidepressant medications (duloxetine, escitalopram, sertraline, or venlafaxine extended release [XR]) on Day 1 that will be continued for the duration of the 4-week Double-Blind Treatment Phase.
  Interventions: Drug: Esketamine 56 mg; Drug: Esketamine 84 mg; Drug: Duloxetine (Oral Antidepressant); Drug: Escitalopram (Oral Antidepressant); Drug: Sertraline (Oral Antidepressant); Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant)
- Oral Antidepressant plus Intranasal Placebo (Active Comparator): Eligible Participants will self-administer matching placebo intranasally twice per week for 4 weeks in Double-Blind Treatment Phase. In addition, participants will simultaneously initiate a new, open-label oral antidepressant medications (duloxetine, escitalopram, sertraline, or venlafaxine XR) on Day 1 that will be continued for the duration of Double-Blind Treatment Phase.
  Interventions: Drug: Placebo; Drug: Duloxetine (Oral Antidepressant); Drug: Escitalopram (Oral Antidepressant); Drug: Sertraline (Oral Antidepressant); Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant)

INTERVENTIONS:
Drug: Esketamine 56 mg — Participants will self-administer 56 mg of esketamine as intranasal spray.
  Arms: Intranasal Esketamine plus Oral Antidepressant
Drug: Esketamine 84 mg — Participants will self-administer 84 mg of esketamine as intranasal spray.
  Arms: Intranasal Esketamine plus Oral Antidepressant
Drug: Placebo — Participants will self-administer matching placebo as intranasal spray.
  Arms: Oral Antidepressant plus Intranasal Placebo
Drug: Duloxetine (Oral Antidepressant) — Duloxetine can be selected as the oral antidepressant medication based on investigator's discretion. The minimum therapeutic dose is 60 milligram per day (mg/day).
Drug: Escitalopram (Oral Antidepressant) — Escitalopram can be selected as the oral antidepressant medication based on investigator's discretion. Escitalopram will be started at a dose of 10 mg/day and up-titrated to a maximum dose of 20 mg/day.
Drug: Sertraline (Oral Antidepressant) — Sertraline can be selected as the oral antidepressant medication based on investigator's discretion. Sertraline will be started at a dose of 50 mg/day and up-titrated to a maximum dose of 200 mg/day.
Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant) — Venlafaxine XR can be selected as the oral antidepressant medication based on investigator's discretion. Venlafaxine XR will be started at a dose of 75 mg/day and up-titrated to a maximum dose of 225 mg/day.

SUMMARY:
The purpose of this study is to evaluate the efficacy of switching adult participants with treatment-resistant depression (TRD) from a prior antidepressant treatment (to which they have not responded) to flexibly dosed intranasal esketamine (56 milligram [mg] or 84 mg) plus a newly initiated oral antidepressant compared with switching to a newly initiated oral antidepressant (active comparator) plus intranasal placebo, in improving depressive symptoms. Efficacy will be assessed by the change from baseline in the Montgomery Asberg Depression Rating Scale (MADRS) total score from Day 1 (before randomization) to the end of the 4-week double-blind treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* At the start of the screening/prospective observational phase, participant must meet the Diagnostic and Statistical Manual of Mental Disorders-fifth edition (DSM-5) diagnostic criteria for recurrent major depressive disorder (MDD) or single-episode MDD, without psychotic features, based upon clinical assessment and confirmed by the Mini-International Neuropsychiatric Interview (mental status questionnaire) (MINI)
* At the start of the screening/prospective observational phase, participant must have had non-response (less than or equal to [<=] 25 percent [%] improvement) to >=1 but <=5 (if current episode is greater than (>) 2 years or not definable, upper limit is applicable to only the last 2 years) oral antidepressant treatments in the current episode of depression, assessed using the Massachusetts General Hospital - Antidepressant Treatment Response Questionnaire (MGH-ATRQ) and confirmed by documented records (for example, medical/ pharmacy/prescription records or letter from a treating physician). In addition, the participant is taking a different oral antidepressant treatment (on the MGH-ATRQ) for at least the previous 2 weeks at or above the minimum therapeutic dose
* The participant's current major depressive episode, depression symptom severity (Week 1 Montgomery-Asberg Depression Rating Scale [MADRS] total score >=28 required), and antidepressant treatment response in the current depressive episode, must be confirmed using a Clinical-Validation Inventory for Study Admission (C-VISA)
* Participant must be medically stable on the basis of physical examination, medical history, vital signs (including blood pressure), pulse oximetry, and 12-lead electrocardiogram (ECG) performed in the screening/prospective observational phase. If there are any abnormalities that are not specified in the inclusion and exclusion criteria, they must be consistent with the underlying illness in the study population. This determination must be recorded in the participant's source documents and initialed or signed by the investigator
* Participant must be medically stable on the basis of clinical laboratory tests performed in the screening/prospective observational phase. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed or signed by the investigator

Exclusion Criteria:

* The participant's depressive symptoms have previously demonstrated non-response to:

  1. Esketamine or ketamine in the current major depressive episode per clinical judgment, or
  2. All of the oral antidepressant treatment options available in the respective country for the double-blind phase (that is, duloxetine, escitalopram, sertraline, and venlafaxine XR) in the current major depressive episode (based on MGH-ATRQ), or
  3. An adequate course of treatment with electroconvulsive therapy (ECT) in the current major depressive episode, defined as at least 7 treatments with unilateral/bilateral ECT
* Participant has received vagal nerve stimulation (VNS) or has received deep brain stimulation (DBS) in the current episode of depression
* Participant has a current or prior DSM-5 diagnosis of a psychotic disorder or MDD with psychotic features, bipolar or related disorders (confirmed by the MINI), obsessive compulsive disorder (current only), intellectual disability (DSM-5 diagnostic codes 315.8, 317, 318.0, 318.1, 318.2 and 319), autism spectrum disorder, borderline personality disorder, antisocial personality disorder, histrionic personality disorder, or narcissistic personality disorder
* Participant has homicidal ideation/intent, per the investigator's clinical judgment, or has suicidal ideation with some intent to act within 6 months prior to the start of the screening/prospective observational phase, per the investigator's clinical judgment or based on the Columbia Suicide Severity Rating Scale (C-SSRS), corresponding to a response of "Yes" on Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) for suicidal ideation on the C-SSRS, or a history of suicidal behavior within the past year prior to the start of the screening/prospective observational phase. Participants reporting suicidal ideation with intent to act or suicidal behavior prior to the start of the double-blind treatment phase should be excluded
* Participant has a history of moderate or severe substance or alcohol use disorder according to DSM-5 criteria, except nicotine or caffeine, within 6 months before the start of screening/prospective observational phase a. A history (lifetime) of ketamine, phencyclidine (PCP), lysergic acid diethylamide (LSD), or 3, 4-methylenedioxy-methamphetamine (MDMA) hallucinogen-related use disorder is exclusionary

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (30):
- United States (6):
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Biomedical Research Foundation of Northwest Louisiana, Shreveport, Louisiana
  - CBH Health, Gaithersburg, Maryland
  - Adams Clinical, Watertown, Massachusetts
  - The Medical Research Network, LLC, New York, New York
  - IPS Research Company, Oklahoma City, Oklahoma
- China (24):
  - Beijing Anding Hospital of Capital Medical University, Beijing
  - Beijing HuiLong Guan Hospital, Beijing
  - Peking University Sixth Hospital, Beijing
  - The Second People's Hospital of Hunan Province / Brian Hospital of Hunan Province, Changsha
  - The second Xiangya Hospital of Central South University, Changsha
  - West China Hospital Sichuan University, Chengdu
  - Chongqing Mental Health Center, Chongqing
  - the 3rd Affiliated Hospital,Sun Yansen University, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Hangzhou Seventh People's Hospital, Hangzhou
  - First Hospital, Zhejiang University Medical College, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou
  - Huzhou third people's Hospital, Huzhou
  - First Affiliated Hospital of Kunming Medical Unversity, Kunming
  - Nanjing Brain Hospital Affilicated to Nanjing Medical University, Nanjing
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Anding Hospital, Tianjin
  - Urumqi fourth Hospital, Ürümqi
  - The first affiliated hospital of Xinjiang medical university, Ürümqi
  - Renmin Hospital of Wuhan University, Wuhan
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - Xi'an Mental Health Center, Xi'an
  - Xiamen Xianyue Hospital, Xiamen
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

RESULTS

PARTICIPANT FLOW:
Groups:
- Intranasal Esketamine + Oral Antidepressant (AD): Participants received intranasal esketamine 56 milligrams (mg) or 84 mg twice per week for 4 weeks as a flexible dose regimen. All participants started at a dose of 56 mg on Day 1. The dose could be increased to 84 mg or maintained at 56 mg per investigator's discretion. Participants simultaneously received 1 of the 4 open-label oral antidepressant treatment (duloxetine, escitalopram, sertraline, or venlafaxine extended release [XR]) on Day 1 that was continued for the duration of the 4-week Double-Blind Treatment Phase. The follow-up phase included participants who received at least 1 dose of intranasal study medication in the double-blind treatment phase. Participants received oral AD for 8 weeks in the follow-up phase unless it was determined not to be clinically appropriate.
- Intranasal Placebo + Oral AD: Participants received intranasal placebo twice per week for 4 weeks as a flexible dose regimen. Participants simultaneously received 1 of the 4 open-label oral antidepressant treatment (duloxetine, escitalopram, sertraline, or venlafaxine XR) on Day 1 that was continued for the duration of the 4-week Double-Blind Treatment Phase. The follow-up phase included participants who received at least 1 dose of intranasal study medication in the double-blind treatment phase. Participants received oral AD for 8 weeks in the follow-up phase unless it was determined not to be clinically appropriate.
Period: Double Blind Treatment Phase (4 Weeks)
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Started | 126 | 126
Full Analysis Set | 124 | 126
Completed | 108 | 106
Not Completed | 18 | 20
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lack of Efficacy | 3 | 14
Not completed — Adverse Event | 7 | 2
Not completed — Death | 1 | 0
Not completed — Covid-19 related | 2 | 2
Not completed — Non-compliance with study drug | 0 | 1
Not completed — Other | 2 | 0
Period: Follow-up Phase (Up to 8 Weeks)
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Started | 106 | 103
Completed | 99 | 100
Not Completed | 7 | 3
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Investigator decision to discontinue follow-up and proceed to 54135419TRD3008 (NCT02782104) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD | Total
Number analyzed (Participants) | 126 | 126 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 126 | 126 | 252
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (11.95) | 37.8 (12.36) | 37.3 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 55 | 113
  Male | 68 | 71 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 121 | 124 | 245
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 112 | 112 | 224
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 12 | 9 | 21
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  CHINA | 112 | 112 | 224
  UNITED STATES | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score to the End of Double-blind Treatment Phase (Day 28)
Description: The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, inability to feel (interest level), pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), summed for a total possible score range of 0 to 60. Higher scores represent a more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline up to end of the double-blind treatment phase (Day 28)
Population: Full analysis set included all randomized participants who received a least 1 dose of intranasal study medication and 1 dose of oral antidepressant medication during the double-blind treatment phase. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Number analyzed (Participants) | 109 | 106
Units on a Scale | -10.1 (10.80) | -8.1 (10.26)
Statistical Analysis 1: Comparison: Intranasal Esketamine + Oral Antidepressant (AD); Test type: Superiority; p = 0.123, Mixed-effects Model for Repeated Measure — 2-sided; Difference of Least Square (LS) Means = -2.0, 95% CI 2-sided [-4.64 to 0.55]

2. Secondary Outcome: Change From Baseline in Depressive Symptoms as Measured by the MADRS Total Score to 24 Hours Post First Dose (Day 2)
Description: as for outcome 1
Time Frame: Baseline (Day 1: predose) to 24 hours post first dose (Day 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Number analyzed (Participants) | 123 | 125
Units on a Scale | -8.0 (9.01) | -4.4 (7.66)
Statistical Analysis 1: Comparison: Intranasal Esketamine + Oral Antidepressant (AD); Test type: Superiority; Difference of LS Means = -3.3, 95% CI 2-sided [-5.33 to -1.33]

3. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score to the End of Double-blind Treatment Phase (Day 28)
Description: The SDS is a subject-reported outcome measure that consists of a 5-item questionnaire which has been widely used and accepted for assessment of functional impairment and associated disability. The first three items assess disruption of (1) work/school, (2) social life, and (3) family life/home responsibilities using a 0-10 rating scale. The score for the first three items are summed to create a total score of 0-30, where a higher score indicates greater impairment. It also has one item on days lost from school or work and one item on days when underproductive.
Time Frame: Baseline up to end of the double-blind treatment phase (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Number analyzed (Participants) | 99 | 98
Units on a Scale | -6.3 (7.54) | -5.3 (7.03)
Statistical Analysis 1: Comparison: Intranasal Esketamine + Oral Antidepressant (AD); Test type: Superiority; Difference of LS Means = -1.0, 95% CI 2-sided [-2.96 to 0.97]

4. Secondary Outcome: Percentage of Participants With Onset of Clinical Response
Description: Onset of clinical response is defined as greater than or equal to (>=) 50 percent (%) improvement from baseline in MADRS total score with onset by Day 2 that was maintained through Day 28. The MADRS scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, inability to feel (interest level), pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), summed for a total possible score range of 0 to 60. Higher scores represent a more severe condition. Negative change in score indicates improvement.
Time Frame: Day 2 up to Day 28
Population: Full analysis set included all randomized participants who received a least 1 dose of intranasal study medication and 1 dose of oral antidepressant medication during the double-blind treatment phase.
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Number analyzed (Participants) | 124 | 126
Percentage of participants | 6.5 | 1.6

5. Secondary Outcome: Percentage of Responders at the End of Double-blind Treatment Phase (Day 28)
Description: Percentage of responders at the end of double-blind treatment phase (Day 28) were assessed. A participant was defined as a responder at a given time point if the percent improvement from baseline in MADRS total score is at least 50%. The MADRS scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, inability to feel (interest level), pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), summed for a total possible score range of 0 to 60. Higher scores represent a more severe condition. Negative change in score indicates improvement.
Time Frame: Day 28
Population: as for outcome 1
Measure: Number; unit: Percentage of Responders
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Number analyzed (Participants) | 109 | 106
Percentage of Responders | 19.3 | 16.0

6. Secondary Outcome: Percentage of Participants in Remission at the End of Double-blind Treatment Phase (Day 28)
Description: Percentage of participants in remission at the end of double-blind treatment phase (Day 28) were assessed. A participant was considered as a remitter if participant had a MADRS total score of less than or equal to [<=] 12 at a visit. MADRS scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, inability to feel (interest level), pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), summed for a total possible score range of 0 to 60. Higher scores represent a more severe condition. Negative change in score indicates improvement.
Time Frame: Day 28
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Number analyzed (Participants) | 109 | 106
Percentage of Participants | 12.8 | 10.4

7. Secondary Outcome: Percentage of Participants With Sustained Remission
Description: Sustained remission is defined as the first occurrence of remission (MADRS Total score <=12) that was maintained through the Day 28 assessment with one excursion prior to Day 28. The MADRS scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, inability to feel (interest level), pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), summed for a total possible score range of 0 to 60. Higher scores represent a more severe condition. Negative change in score indicates improvement.
Time Frame: Up to Day 28
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Number analyzed (Participants) | 124 | 126
Percentage of Participants | 5.6 | 6.3

8. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity (CGI-S) Scale Score up to the Endpoint (Double-blind Treatment Phase [Day 28])
Description: The CGI-S provides an overall clinician-determined summary measure of the severity of the participant's illness that takes into account all available information, including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. The CGI-S evaluates the severity of psychopathology on a scale of 1 to 7. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating according to: 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. The CGI-S permits a global evaluation of the participant's condition at a given time. Negative change in score indicates improvement. The last post-baseline observation during the double-blind phase was carried forward as Endpoint.
Time Frame: Baseline up to Double-blind Endpoint (Day 28)
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Number analyzed (Participants) | 121 | 126
Units on a Scale | -1.0 [-5 to 1] | -1.0 [-5 to 1]

9. Secondary Outcome: Change From Baseline in Generalized Anxiety Disorder 7-item (GAD-7) Scale Score up to the Endpoint (Double-blind Treatment Phase [Day 28])
Description: The GAD-7 is a brief and validated 7-item self-reported assessment of overall anxiety. Participants respond to each item using a 4 point scale with response categories of 0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day. Item responses are summed to yield a total score with a range of 0 to 21, where higher scores indicate more anxiety. The recall period is 2 weeks. The severity of the GAD-7 is categorized as follows: None (0-4), Mild (5-9), Moderate (10-14) and Severe (15-21). The last post-baseline observation during the double-blind phase was carried forward as the "Endpoint".
Time Frame: Baseline up to Endpoint (double-blind treatment phase [Day 28])
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Number analyzed (Participants) | 118 | 120
Units on a Scale | -4.3 (5.65) | -2.9 (5.28)

10. Secondary Outcome: Change From Baseline in Participant-Reported Health-Related Quality of Life as Assessed by EuroQol-5 Dimension-5 Level (EQ-5D-5L) Score up to the Endpoint (Double-blind Treatment Phase [Day 28]): Health Status Index
Description: The EQ-5D-5L is a standardized 2-part instrument for use as a measure of health outcome, primarily designed for self-completion by respondents. It essentially consists of the EQ-5D-5L descriptive system and the EQ Visual Analogue Scale (EQ-VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of the 5 dimensions is divided into 5 levels of perceived problems (Level 1 indicating no problem, Level 2 indicating slight problems, Level 3 indicating moderate problems, Level 4 indicating severe problems, and Level 5 indicating extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a HSI. Health Status Index ranges from -0.148 to 0.949, and is anchored at 0 (dead) and 1 (full health), a lower score indicates worse health.
Time Frame: Baseline up to Double-blind Endpoint (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Number analyzed (Participants) | 120 | 123
Units on a Scale | 0.152 (0.2294) | 0.103 (0.2084)

11. Secondary Outcome: Change From Baseline in Participant-Reported Health Status as Assessed by EuroQol-5 Dimension-5 Level (EQ-5D-5L) Score up to the Endpoint (Double-blind Treatment Phase [Day 28]): Visual Analogue Scale (VAS)
Description: The EQ-5D-5L is a standardized 2-part instrument for use as a measure of health outcome, primarily designed for self-completion by respondents. It essentially consists of the EQ-5D-5L descriptive system and the EQ-VAS. EQ-VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Positive change in score indicates improvement.
Time Frame: Baseline up to Double-blind Endpoint (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Number analyzed (Participants) | 120 | 123
Units on a Scale | 16.7 (20.47) | 11.9 (25.21)

12. Secondary Outcome: Change From Baseline in Participant-Reported Health Status as Assessed by EuroQol-5 Dimension-5 Level (EQ-5D-5L) up to the Endpoint (Double-blind Treatment Phase [Day 28]): Sum Score
Description: EQ-5D-5L consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ-VAS). EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a Health Status Index (HSI). HSI ranges from -0.148 to 0.949 and is anchored at 0 (health state value equal to dead) and 1 (full health). EQ-VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Sum score ranges from 0 to 100 where, sum score = (sum of the scores from the 5 dimensions minus 5) *5. Higher score indicates worst health state.
Time Frame: Baseline up to Double-blind Endpoint (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant (AD) | Intranasal Placebo + Oral AD
Number analyzed (Participants) | 120 | 123
Units on a Scale | -13.4 (18.83) | -9.5 (16.95)

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Description: The safety analysis set (SAS) included all randomized participants who received at least 1 dose of intranasal study medication or 1 dose of oral antidepressant medication during the double-blind treatment phase. The Follow-up analysis set included all subjects who entered the follow-up phase. Safety analysis was done on SAS for double-blind phase and Follow-up analysis set for follow-up phase.
Groups:
- Double-blind: Intranasal Esketamine+ Oral Antidepressant (AD): Participants received intranasal esketamine 56 milligrams (mg) or 84 mg twice per week for 4 weeks as a flexible dose regimen. All participants started at a dose of 56 mg on Day 1. The dose could be increased to 84 mg or maintained at 56 mg per investigator's discretion. Participants simultaneously received 1 of the 4 open-label oral antidepressant treatment (duloxetine, escitalopram, sertraline, or venlafaxine extended release [XR]) on Day 1 that was continued for the duration of the 4-week Double-Blind Treatment Phase.
- Double-blind: Oral AD + Intranasal Placebo: Participants received intranasal placebo twice per week for 4 weeks as a flexible dose regimen. Participants simultaneously received 1 of the 4 open-label oral antidepressant treatment (duloxetine, escitalopram, sertraline, or venlafaxine XR) on Day 1 that was continued for the duration of the 4-week Double-Blind Treatment Phase.
- Follow-up: Intranasal Esketamine+ Oral AD; Follow-up: Oral AD + Intranasal Placebo: The follow-up phase included participants who received at least 1 dose of intranasal study medication in the double-blind treatment phase. Participants received oral AD for 8 weeks of the follow-up phase unless it was determined to not be clinically appropriate. No intranasal study medication was administered during this phase.
Arm/Group | Double-blind: Intranasal Esketamine+ Oral Antidepressant (AD) | Double-blind: Oral AD + Intranasal Placebo | Follow-up: Intranasal Esketamine+ Oral AD | Follow-up: Oral AD + Intranasal Placebo
All-Cause Mortality (participants affected / at risk) | 1/126 | 0/126 | 0/106 | 0/103
Serious Adverse Events (participants affected / at risk) | 3/126 | 3/126 | 2/106 | 2/103
Other Adverse Events (participants affected / at risk) | 118/126 | 61/126 | 10/106 | 13/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind: Intranasal Esketamine+ Oral Antidepressant (AD) (N=126) | Double-blind: Oral AD + Intranasal Placebo (N=126) | Follow-up: Intranasal Esketamine+ Oral AD (N=106) | Follow-up: Oral AD + Intranasal Placebo (N=103)
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Completed Suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 3 | 1 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind: Intranasal Esketamine+ Oral Antidepressant (AD) (N=126) | Double-blind: Oral AD + Intranasal Placebo (N=126) | Follow-up: Intranasal Esketamine+ Oral AD (N=106) | Follow-up: Oral AD + Intranasal Placebo (N=103)
Vision Blurred (Eye disorders) | 23 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 1 | 6
Hypoaesthesia Oral (Gastrointestinal disorders) | 10 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 53 | 17 | 0 | 3
Vomiting (Gastrointestinal disorders) | 23 | 2 | 0 | 2
Asthenia (General disorders) | 8 | 2 | 1 | 0
Fatigue (General disorders) | 8 | 7 | 1 | 0
Feeling Drunk (General disorders) | 11 | 2 | 0 | 0
Blood Pressure Increased (Investigations) | 38 | 13 | 1 | 2
Dizziness (Nervous system disorders) | 97 | 25 | 0 | 1
Dysgeusia (Nervous system disorders) | 14 | 6 | 0 | 1
Headache (Nervous system disorders) | 16 | 14 | 3 | 0
Hypoaesthesia (Nervous system disorders) | 25 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 20 | 11 | 0 | 1
Anxiety (Psychiatric disorders) | 8 | 3 | 2 | 0
Dissociation (Psychiatric disorders) | 75 | 8 | 0 | 1
Euphoric Mood (Psychiatric disorders) | 9 | 1 | 0 | 0
Hallucination, Visual (Psychiatric disorders) | 7 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 7 | 11 | 3 | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
As esketamine has known transient dissociative effects that are difficult to blind, these specific treatment-emergent events could have biased the staff who provided and observed the dosing. Therefore, to ensure an unbiased efficacy evaluation, independent, remote (by telephone), blinded MADRS raters were used to assess the treatment response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT03434041/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT03434041/SAP_001.pdf